CLINICAL TRIAL: NCT06658795
Title: Effects of Transcranial Direct Current Stimulation on Loneliness in Older Adults With Depression: A Randomized Controlled Trial
Brief Title: Treating Loneliness In The Older Adult With Depression With tDCS
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Guangzhou Psychiatric Hospital (Other Government)
Collaborators: The University of Hong Kong (Other)
Responsible Party: Principal Investigator, Kangguang Lin, Director of the Department of Affective disorders, Guangzhou Psychiatric Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 2024-17
Record Dates: First submitted 2024-10-22; First posted 2024-10-26 (Actual); Last update posted 2024-10-26 (Actual); Status verified 2024-10

CONDITIONS: Major Depressive Disorder; Loneliness
Keywords: Randomization Controlled Trial; Transcranial Direct Current Stimulation; Depression; loneliness
MeSH Terms: conditions — Depressive Disorder, Major; Depression | interventions — Transcranial Direct Current Stimulation

STUDY DESIGN:
Intervention Model Description: The tDCS parameters were set to a current of 2mA for a single session lasting 20 minutes. Based on the EEG 10-20 international system, the positive electrode for stimulating the rVLPFC was placed at position F6, while the negative electrode was placed in the left supraorbital area/FP1 (e.g., He et al., 2020, Psychol Med) (Figure 1-5a). For stimulating the lDLPFC, the positive electrode was placed at position F3, and the negative electrode was placed in the right supraorbital area/FP2 (e.g., Dubreuil-Vall et al., 2021, Biol Psychiatry: CNNI) (Figure 1-5b). In the sham stimulation group, the electrode positions were randomized to match those of the rVLPFC or lDLPFC groups, but the stimulation only lasted for the first 30 seconds.
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Left DLPFC stimulation group (Experimental): The tDCS parameters were set to a current of 2mA for a single session lasting 20 minutes. Based on the EEG 10-20 international system, the positive electrode was placed at position F3, and the negative electrode was placed in the right supraorbital area/FP2 (e.g., Dubreuil-Vall et al., 2021, Biol Psychiatry: CNNI)
  Interventions: Device: Transcranial direct current stimulation (tDCS) on the Left DLPFC
- Right VLPFC stimulation group (Experimental): The tDCS parameters were set to a current of 2mA for a single session lasting 20 minutes. Based on the EEG 10-20 international system, the positive electrode for stimulating the right VLPFC was placed at position F6, while the negative electrode was placed in the left supraorbital area/FP1 (e.g., He et al., 2020, Psychol Med).
  Interventions: Device: Transcranial direct current stimulation (tDCS) on the right VLPFC
- Sham stimulation group (Sham Comparator): In the sham stimulation group, the electrode positions were randomized to match those of the rVLPFC or lDLPFC groups, but the stimulation only lasted for the first 30 seconds.
  Interventions: Device: Sham stimulation group

INTERVENTIONS:
Device: Transcranial direct current stimulation (tDCS) on the Left DLPFC — The tDCS parameters were set to a current of 2mA for a single session lasting 20 minutes. For stimulating the lDLPFC, the positive electrode was placed at position F3, and the negative electrode was placed in the right supraorbital area/FP2 (e.g., Dubreuil-Vall et al., 2021, Biol Psychiatry: CNNI).
  Arms: Left DLPFC stimulation group
Device: Transcranial direct current stimulation (tDCS) on the right VLPFC — The tDCS parameters were set to a current of 2mA for a single session lasting 20 minutes. Based on the EEG 10-20 international system, the positive electrode for stimulating the rVLPFC was placed at position F6, while the negative electrode was placed in the left supraorbital area/FP1 (e.g., He et al., 2020, Psychol Med)
  Arms: Right VLPFC stimulation group
Device: Sham stimulation group — The electrode positions were randomized to match those of the rVLPFC or lDLPFC groups, but the stimulation only lasted for the first 30 seconds.
  Arms: Sham stimulation group

SUMMARY:
High loneliness is prevalent among older adults and is a significant risk factor for major depression and low recovery rates in patients. Current interventions for loneliness are limited. Previous research has demonstrated a link between loneliness, negative social emotions, and reduced resting-state functional connectivity in the lateral prefrontal cortex (LPFC) and the default mode network (DMN). Transcranial direct current stimulation (tDCS) has shown promise in enhancing emotional regulation and connectivity, potentially alleviating loneliness in older adults with depression.

DETAILED DESCRIPTION:
Loneliness is a pervasive issue among older adults, significantly increasing the risk of major depression and contributing to low recovery rates in affected individuals. Despite its widespread impact, current interventions aimed at alleviating loneliness remain limited and often ineffective. Research has revealed a strong connection between feelings of loneliness, negative social emotions, and decreased resting-state functional connectivity in key brain regions, particularly the lateral prefrontal cortex (LPFC) and the default mode network (DMN). These findings suggest that the neural underpinnings of loneliness may be targeted to improve emotional well-being.

Transcranial direct current stimulation (tDCS) emerges as a promising intervention in this context, as it has been shown to enhance emotional regulation and improve functional connectivity within these neural networks. By applying low electrical currents to specific brain areas, tDCS may help mitigate feelings of loneliness, thereby fostering a greater sense of social connection among older adults with depression.

Objectives Evaluate the Effects of Repeated tDCS on Loneliness Levels: This trial aims to systematically assess how repeated sessions of tDCS influence loneliness in older adults with major depressive disorder. By comparing these groups, we hope to understand the differential impacts of tDCS on loneliness, taking into account the potential confounding effects of depression.

Elucidate the Neuro-Emotional Mechanisms: A key objective is to uncover the neuro-emotional mechanisms that underlie the effects of tDCS on loneliness. This involves examining changes in neural activity and connectivity patterns in the LPFC and DMN, as well as tracking shifts in negative social emotions that may accompany improvements in loneliness. Understanding these mechanisms could enhance the efficacy of tDCS as an intervention.

Develop Predictive Models for Individualized Treatment Outcomes: Another important aim of this trial is to create predictive models that utilize neuro-emotional data to tailor treatment approaches for individuals. By identifying specific neural and emotional markers that correlate with positive outcomes from tDCS, we can move toward more personalized interventions, potentially improving recovery rates and overall mental health in older adults with depression facing loneliness.

This trial represents a significant step toward addressing the critical issue of loneliness in older adults with depression, with the potential to offer a novel and effective intervention strategy that integrates neurobiology and emotional health.

ELIGIBILITY:
Inclusion Criteria:

* High loneliness (UCLA Loneliness Scale > 43).
* Diagnosis of major depressive disorder confirmed by the Structured Clinical Interview for DSM-5 Disorders.
* absence of suicidal ideation (Hamilton Depression Scale item 3 score ≤ 1).

Exclusion Criteria:

* Severe neurological diseases.
* Bipolar disorder, schizophrenia, addiction, or impulse control disorders.
* Contraindications for tDCS or MRI (e.g., metal implants).
* Presence of suicidal ideation.

Ages: 60 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — Participant eligibility is based on self-representation of gender identity.
Enrollment: 180 (Estimated)
Dates: Start 2024-10-29 (Estimated); Primary Completion 2026-10-20 (Estimated); Study Completion 2026-12-30 (Estimated)

PRIMARY OUTCOMES:
Change in loneliness levels from baseline measured by the UCLA Loneliness Scale from baseline | 2 weeks, 1.5 months and 3.5 months
  This outcome measures the change in loneliness levels among participants, assessed using the UCLA Loneliness Scale. Evaluations will occur at baseline, 1 month, and 3 months post-intervention (after the two weeks of intervention, the same as below) to determine the effectiveness of the tDCS intervention on reducing feelings of loneliness in patients with depression.

SECONDARY OUTCOMES:
Change in Emotional and Motivational Ratings from baseline | 2 weeks, 1.5 months and 3.5 months
  Participants' emotional and motivational responses will be assessed using a word rating task, which evaluates how different words or stimuli evoke emotional and motivational reactions.
changes in Social Participation Levels from baseline | 2 weeks, 1.5 months and 3.5 months
  The PM-3D4D questionnaire will be utilized to assess participants' levels of social participation, focusing on engagement in social activities and interactions.
changes in Social Motivation from baseline | 2 weeks, 1.5 months and 3.5 months
  Social motivation will be evaluated through the Social Motivation Questionnaire, which examines the intrinsic and extrinsic factors that drive social engagement in individuals.
changes in Social Network from baseline | 2 weeks, 1.5 months and 3.5 months
  The Lubben Social Network Scale will be used to assess participants' social networks
changes in Emotional Regulation from baseline | 2 weeks, 1.5 months and 3.5 months
  The Cognitive Emotion Regulation Questionnaire will be used to assess participants' emotion regulation functions.
changes in Affective Traits from baseline | 2 weeks, 1.5 months and 3.5 months
  Affective traits will be evaluated using the Chinese Affect Scale, which assess individual differences in emotional experiences and behavioral tendencies.
changes in Reward Sensitivity from baseline | 2 weeks, 1.5 months and 3.5 months
  The Temporal Experience of Pleasure Scale will be used to assess participants' reward sensitivity.
changes in Depressive Symptoms from baseline | 2 weeks, 1.5 months and 3.5 months
  Hamilton Depression Rating Scale (HAM-D) will be employed to measure the severity of depressive symptoms among participants, providing insight into their mental health status.
changes in Resting-State Functional Connectivity from baseline | 2 weeks, 1.5 months and 3.5 months
  Resting State Functional Connectivity among major brain networks based on T2-weighted functional magnetic resonance imaging data will be assessed.
Change in social support from baseline | 2 weeks, 1.5 months and 3.5 months
  the Multidimensional Scale of Perceived Social Support will be used to assess participants' perceived social support
changes in Emotion Coping from baseline | 2 weeks, 1.5 months and 3.5 months
  The COPE questionnaire will be used to assess participants' emotion coping under adversity.
changes in Incentive-Driven Behavioural Tendencies from baseline | 2 weeks, 1.5 months and 3.5 months
  The Behavioural Activation/Inhibition Scale will be used to assess participants' behavioural tendencies driven by rewards and punishments.
changes in Anhedonia level from baseline | 2 weeks, 1.5 months and 3.5 months
  The Dimensional Anhedonia Rating Scale will be used to assess participants' anhedonia level.

CONTACTS AND LOCATIONS:
Locations (1):
- Guangzhou Brain Hospital, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dubreuil-Vall L, Gomez-Bernal F, Villegas AC, Cirillo P, Surman C, Ruffini G, Widge AS, Camprodon JA. Transcranial Direct Current Stimulation to the Left Dorsolateral Prefrontal Cortex Improves Cognitive Control in Patients With Attention-Deficit/Hyperactivity Disorder: A Randomized Behavioral and Neurophysiological Study. Biol Psychiatry Cogn Neurosci Neuroimaging. 2021 Apr;6(4):439-448. doi: 10.1016/j.bpsc.2020.11.006. Epub 2020 Nov 25. PMID 33549516
- [Background] He Z, Liu Z, Zhao J, Elliott R, Zhang D. Improving emotion regulation of social exclusion in depression-prone individuals: a tDCS study targeting right VLPFC. Psychol Med. 2020 Dec;50(16):2768-2779. doi: 10.1017/S0033291719002915. Epub 2019 Oct 16. PMID 31615594